CLINICAL TRIAL: NCT04162106
Title: Open Label, Single Center, Randomized Study Evaluating the Feasibility of the Ultravision™ Visual Field Clearing System in Low Pressure Laparoscopic Cholecystectomy Compared To AirsealL® IFS
Brief Title: Feasibility of the Ultravision™ System in Low Pressure Laparoscopic Cholecystectomy Compared to Airseal® IFS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alesi Surgical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00103233
Record Dates: First submitted 2019-11-11; First posted 2019-11-14 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Laparoscopic Cholecystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Ultravision™ System (Active Comparator): Smoke management during laparoscopic cholecystectomy performed with the Ultravision™ System
  Interventions: Device: Smoke management during laparoscopic cholecystectomy using the Ultravision™ System
- Airseal® iFS (Active Comparator): Smoke management during laparoscopic cholecsystectomy performed with the Airseal® iFS
  Interventions: Device: Smoke management during laparoscopic cholecystectomy using the Airseal® iFS

INTERVENTIONS:
Device: Smoke management during laparoscopic cholecystectomy using the Ultravision™ System — The Ultravision™ System will be used during the procedure to manage smoke generated as a result of the use of diathermy.
  Arms: Ultravision™ System
Device: Smoke management during laparoscopic cholecystectomy using the Airseal® iFS — The Airseal® iFS will be used during the procedure to manage smoke generated as a result of the use of diathermy.
  Arms: Airseal® iFS

SUMMARY:
This post-market clinical study is designed to evaluate the effectiveness of the Ultravision™ System when compared to the Airseal® iFS within an approved indication for use, namely laparoscopic cholosystectomy.

DETAILED DESCRIPTION:
The primary hypothesis being tested in this study is that Ultravision facilitates the utilization of lower pneumoperitoneal pressures whilst maintaining an adequate visual field throughout the procedure with low demand for CO2 replenishment to maintain pneumoperitoneal pressure. Comparisons in terms of surgical field visualization, procedure times, and CO2 consumption will be conducted in order to determine whether or not any clinical benefits are derived from the use of the Ultravision™ System compared to the Airseal® iFS. Low pressure laparoscopy for this study is set at 10mmHg. This is a prospective, open-label, randomized controlled study. The study will include two study arms. Patients undergoing laparoscopic cholecystectomy will be randomized to either "Ultravision" (study arm 1) or Airseal® iFS (study arm 2). Both groups will conduct the procedure at 10mmHg, considered to be low pressure/low impact laparoscopic surgery. The study will enroll 30 patients, 15 per group. Both devices are being used according to their cleared label claims.

ELIGIBILITY:
Inclusion Criteria:

* Is 18 years or older
* Provide written informed consent prior to trial procedures after studies indicate that the patient needs the prescribed procedure
* Agrees to attend all follow-up assessments
* Is indicated for elective laparoscopic cholecystectomy

Exclusion Criteria:

* Existing comorbidities that would contraindicate them for laparoscopic surgery
* Patient anatomy i.e. abdominal wall thickness that exceeds the working length of the Ionwand catheter identified intraoperatively
* Body Mass Index > 50
* Be pregnant (if female)
* Has a condition of unrelated chronic pain requiring medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Carbon Dioxide Utilization | Measured from Veress needle insertion to just prior to gall bladder removal
  The volume measured in Liters of Carbon Dioxide consumed during the procedure
Quality of Visualization | Measured from camera insertion through removal
  The quality of visualization in the laparoscopic field

SECONDARY OUTCOMES:
Procedure time for Diathermy use | Measured from the exposure and identification of the cystic duct and artery is complete to the last use of diathermy
  Measures the procedure time in minutes where diathermy is used
Diathermy Power Setting | Measured from the exposure and identification of the cystic duct and artery is complete to the last use of diathermy
  Highest diathermy setting used during the procedure
Procedure Time | Measured from the insertion of the camera to the time of closure
  Overall procedure time in minutes
End tidal CO2 Volume | Measured at Veress needle insertion and just prior to gall bladder removal
  End tidal volume of CO2
Laparoscope cleaning | Measured from the exposure and identification of the cystic duct and artery is complete to the last use of diathermy
  The number of times during the procedure that the laparoscope must be removed for cleaning to maintain visual field
Pneumoperitoneum Pressure | Starting pneumoperitoneum pressure at the time of camera trocar insertion, record the maximum pressure that occurred during the procedure
  The pneumoperitoneum pressure during the procedure and record of any increase beyond 10mmHg for visualization
Trocar Venting | Measured from the exposure and identification of the cystic duct and artery is complete to the last use of diathermy
  The number of times the trocar is used to vent during the procedure for visualization
Case Complexity | Immediately post-procedure
  Case complexity compared to surgeon experience. Recorded as simple or routine or complex/difficult.
Pain Assessment | Pre-procedure and 1 to 7 days post procedure
  Pre and Post operative pain surveys
Pain Medications | 1 to 7 days post procedure
  Amount and type of pain medication administered and record of use following the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Duke Regional Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No